CLINICAL TRIAL: NCT02810769
Title: The Acute Effect of Two Berry Extracts on Cognition and Mood in Adults Aged 40 to 60
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: The New Zealand Institute of Plant and Food Research Ltd. (Other Government)
Responsible Party: Principal Investigator, Anthony Watson, Principal Investigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 28AI5
Record Dates: First submitted 2012-11-08; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Ageing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): Sugar matched control containing no phytochemicals
  Interventions: Dietary Supplement: Control
- Juiced berry drink (Experimental): Cold pressed berry drink standardised to contain 500mg of berry polyphenols
  Interventions: Dietary Supplement: Berry drink
- Powdered berry drink (Experimental): Berry drink made up from a powdered concentrate. each drink will be standardised to contain 500mg of polyphenols
  Interventions: Dietary Supplement: Powdered berry drink

INTERVENTIONS:
Dietary Supplement: Berry drink — Cold pressed berry drink standardised to contain 500mg of berry polyphenols
  Arms: Juiced berry drink
Dietary Supplement: Control — Sugar matched control containing berry flavouring and no phytochemicals
  Arms: Control
Dietary Supplement: Powdered berry drink — Berry drink made from a powder concentrate standardised to contain 500mg of polyphenols
  Arms: Powdered berry drink

SUMMARY:
The first study of my PhD showed that acute supplementation of berry extracts can modulate cognitive behaviour in healthy adults. There is a growing body of evidence supporting an improvement in memory and learning performance in animal models following the ingestion of flavonoid rich fruits (Shukitt-Hale et al 2008;Spencer 2008; Spencer et al., 2008). However, study 2, showed no effect on any aspects of memory in healthy young adults after supplementation of the berry extracts. It is hypothesised that the lack of behavioural effects on memory of the berry juice in study 2 was because of the cohort used. These healthy adult participants were already performing near to their peak (Salthouse et al., 2009), and unlike study one, participants were not mentally fatigued enough to reveal subtle cognitive benefits.

The aims of the study are to examine if acute supplementation of two berry extracts in an older population can augment memory, attention and executive function. Secondly, the time course of these behavioural effects will be measured by multiple cognitive assessments throughout the day after consumption of the extracts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smokers
* Aged between 40 and 60 years

Exclusion Criteria:

* History of neurological, vascular or psychiatric illness.
* BMI greater than 35 kg/m2
* Current diagnosis of depression and/or anxiety.
* History or current diagnosis of drug/alcohol abuse.
* Anaemia.
* Any heart disorder.
* Hypertension
* Any respiratory disorder.
* Diabetes.
* Food intolerances/sensitivities.
* Phenylketonuria.
* Use tobacco products or have ceased in the last 6 months.
* Currently taking, or have taken in the last 2 weeks, any prescribed, illicit or herbal drugs and food supplements.
* Any known active infections.
* HIV antibody positive.
* Currently have, have ever had, or may be at risk of hepatitis.
* Have suffered from jaundice within the last year.
* Have haemophilia or any similar clotting disorder.
* History of head trauma
* History of migraines
* History of learning difficulties
* Any Issues with giving blood samples.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Change from baseline at 60, 140, 180, 200, 230 and 350 minutes post dose
Blood lactate | Change from baseline at 60, 140, 180, 200, 230 and 350 minutes post dose
Monoamine oxidase B inhibition | Change from baseline at 350 minutes post dose
Cognitive Measures - Memory- Assessed using a computerised cognitive batter. | Change from baseline 60, 150, 240 and 360 minutes post dose
Cognitive Measures - Attention- Assessed using a computerised cognitive batter. | Change from baseline 60, 150, 240 and 360 minutes post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Brain, Performance and Nutrition Research Centre, Newcastle upon Tyne, Newcastle Upon-Tyne, United Kingdom

REFERENCES:
- See also: Related Info — http://www.nutrition-neuroscience.co.uk/